CLINICAL TRIAL: NCT02768766
Title: Multi-Center Phase Ib Study of Intermittent Dosing of the MEK Inhibitor, Selumetinib, in Patients With Advanced Uveal Melanoma Not Previously Treated With a MEK Inhibitor
Brief Title: Intermittent Selumetinib for Uveal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaheer A. Khan (Other)
Collaborators: AstraZeneca (Industry); Melanoma Research Alliance (Other)
Responsible Party: Sponsor-Investigator, Shaheer A. Khan, Associate Professor of Medicine at the Columbia University Medical Center, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ6999
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Uveal Melanoma
Keywords: MEK inhibitor; Selumetinib; hyd-sulfate AZD6244; Uveal melanoma; Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 100mg.
  Interventions: Drug: Selumetinib, 100mg
- Dose Level 2: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 125mg.
  Interventions: Drug: Selumetinib, 125mg
- Dose Level 3: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 150mg.
  Interventions: Drug: Selumetinib, 150mg
- Dose Level 4: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 175mg.
  Interventions: Drug: Selumetinib, 175mg
- Dose Level 5: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 200mg.
  Interventions: Drug: Selumetinib, 200mg
- Dose Level 6: Selumetinib (Experimental): Subjects will receive selumetinib (hyd-sulfate AZD6244) orally twice a day for three days followed by four days off in four week cycles at a dose of 225mg.
  Interventions: Drug: Selumetinib, 225mg

INTERVENTIONS:
Drug: Selumetinib, 100mg — 100mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 1: Selumetinib
Drug: Selumetinib, 125mg — 125mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 2: Selumetinib
Drug: Selumetinib, 150mg — 150mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 3: Selumetinib
Drug: Selumetinib, 175mg — 175mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 4: Selumetinib
Drug: Selumetinib, 200mg — 200mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 5: Selumetinib
Drug: Selumetinib, 225mg — 225mg, oral capsules, twice daily
  An orally active, small molecule with potential antineoplastic activity. Selumetinib is an ATP-independent inhibitor of mitogen-activated protein kinase kinase (MEK) or MAPK/extracellular-signal-regulated kinase (ERK) kinase) 1 and 2. Inhibition of both MEK1 and 2 by selumetinib prevents the activation of MEK1/2 dependent effector proteins and transcription factors, thereby leading to an inhibition of cellular proliferation in various cancers.
  Other Names: hyd-sulfate AZD6244
  Arms: Dose Level 6: Selumetinib

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, intermittent dosing of the drug Selumetinib will have on subjects with uveal melanoma. Selumetinib is a drug that blocks (or turns off) methyl ethyl ketone (MEK), a protein activated in some uveal melanoma cells. Selumetinib is a MEK inhibitor. Blocking MEK may stop the cancer from growing.

DETAILED DESCRIPTION:
Uveal melanoma (UM) is the most common primary intraocular malignancy in adults, and arises from melanocytes within the choroid plexus of the eye. The development of metastasis is common and occurs in approximately 50% of patients with posterior UM within 15 years of initial diagnosis and treatment. As no effective systemic therapy has yet been identified for this disease, outcomes for metastatic UM are poor with a median survival of 12 months.

There is no FDA approved therapy for patients with advanced UM. Studies have shown that inhibition of the Mitogen-activated protein kinase (MAPK) pathway with the MEK inhibitor selumetinib (hyd-sulfate AZD6244) is an effective therapy for uveal melanoma but despite this treatment, cures are not achieved. Although drugs such as selumetinib have been studied when patients take the treatment every day, research has shown that in some cases, it may be better to use the treatment on an intermittent schedule. Such a strategy may reduce the side effects, allow higher doses of the drug to be used, more completely block the MAPK pathway, and prevent the development of drug resistance mechanisms within the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of metastatic or unresectable uveal melanoma. Note - Documentation of mutation status for uveal melanoma will not be required prospectively given the high rate of GNAQ/11 mutations (>90%) in this population
* Able to provide informed consent prior to initiation of study
* Age ≥ 18 years old
* Measurable indicator lesion by RECIST v1.1
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Karnofsky Performance Status ≥ 60% or Eastern Cooperative Oncology Group (ECOG) ≤2
* Ability to take oral medications
* All clinically significant toxicities from prior therapy must be ≤ grade 1 (with the exception of alopecia)
* Organ and marrow function and laboratory values as follows:

  * Adequate marrow function
  * absolute neutrophil count (ANC) >1500 cells/mm3
  * platelet count >100,000/mm3
  * hemoglobin >9.0g/dL
* Adequate hepatic function

  * Angiotensin Sensitivity Test/alternative (AST/ALT)<2.5x upper limit of normal if no documented liver disease or <5x upper limit of normal if documented liver disease
  * Total bilirubin <1.5X upper limit of normal unless known diagnosis of Gilbert's disease
  * Alkaline phosphatase <2.5x upper limit of normal if no documented liver disease or <6x upper limit of normal if documented liver or bone disease
  * Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Negative pregnancy test (serum or urine) for women of child bearing potential
* The effects of selumetinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 weeks after study discontinuation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of selumetinib administration.

Exclusion Criteria:

* Patients who have had chemotherapy or immunotherapy within 4 weeks or radiation therapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents concurrently. Palliative radiation therapy will be allowed as long as the patient meets all other eligibility criteria.
* Have had recent major surgery within a minimum 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib
* Every effort must be made to avoid the use of a concomitant medication that can prolong the corrected QT (QTc) interval while receiving selumetinib (hyd-sulfate AZD6244). If the patient cannot discontinue medications that prolong QTc interval while receiving selumetinib, close cardiac monitoring should be performed.
* Patients with QTc interval >450 msecs or other factors that increase the risk of QTc prolongation or arrhythmic events (ex. Heart failure, hypokalemia, family history of long QT syndrome) including heart failure that meets New York Heart Association (NYHA) class III and IV definitions (see Appendix A) are excluded.
* Prior or current cardiomyopathy including but not limited to the following: known hypertrophic cardiomyopathy, known arrhythmogenic right ventricular cardiomyopathy, previous moderate or severe impairment of left ventricular systolic function (LVEF <45% on echocardiography or equivalent on MuGA) even if full recovery has occurred.
* Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
* Baseline Left ventricular ejection fraction (LVEF) below the LLN or <55% measured by echocardiography or institution's lower limit of normal (LLN) for MUGA
* Severe valvular heart disease
* Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy
* Acute coronary syndrome within 6 months prior to starting treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because selumetinib may be teratogenic or have abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with selumetinib, breastfeeding should be discontinued if the mother is treated with selumetinib.
* HIV positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with selumetinib.
* Prior treatment with a MEK, Ras or Raf inhibitor
* History of current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED) in the eye unaffected by uveal melanoma; intraocular pressure (IOP) >21mmgHG or uncontrolled glaucoma
* History of interstitial lung disease or pneumonitis
* Patients with known Hepatitis B or C
* Refractory nausea and vomiting, active gastrointestinal disease (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Patients taking vitamin E supplements while on study
* Have known or suspected brain metastases or spinal cord compression, unless the condition has been asymptomatic, has been treated with surgery and / or radiation, and has been stable for at least 4 weeks prior to the first dose of study medication
* Any unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy, except for alopecia
* Have evidence of any other significant clinical disorder or laboratory finding that, as judged by the investigator, makes it undesirable for the patient to participate in the study.
* Patients being actively treated for a secondary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of intermittent selumetinib | Up to 8 weeks
  MTD is defined as the dose associated with a target probability of dose limiting toxicity (DLT) of 25%. DLT will be assessed over the course of first two cycles of treatment (i.e., 8 weeks) for dose selection for subsequent patient treatment initiation.

SECONDARY OUTCOMES:
Number of adverse events (AEs) | Up to 2 years
  Number of AE throughout the study to assess the safety and tolerability of intermittent selumetinib
Number of serious adverse events (SAEs) | Up to 2 years
  Number of SAE throughout the study to assess the safety and tolerability of intermittent selumetinib
Number of subjects with Dose Limiting Toxicity (DLT) | 8 weeks
  Number of subjects with DLT throughout the study to assess the safety and tolerability of intermittent selumetinib. Toxicity was graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v. 4.0). For recurrent adverse events (AEs), the highest reported grade per event per patient was assessed. The DLT observation period was 8 weeks from the initiation of treatment. DLT was defined as any of the following: 1) any serious AE deemed related to the investigational treatment (included grade 1 or 2 ocular toxicity requiring dose reduction); 2) receiving <75% of the planned doses during weeks 1-8; and, 3) death related to the investigational regimen.
Overall Response Rate (ORR) | Up to 2 years
  The overall response rate (ORR) was defined as a confirmed complete response (CR) (Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) or partial response (PR) (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters) according to RECIST 1.1 criteria.
Progression Free Survival (PFS) | Up to 2 years
  PFS measured from date of enrollment until the date of progression or death, whichever occurred first.
Overall Survival (OS) | Up to 2 years
  OS defined as the time from the date of enrollment to the date of death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheer Khan, DO, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvajal RD, Piperno-Neumann S, Kapiteijn E, Chapman PB, Frank S, Joshua AM, Piulats JM, Wolter P, Cocquyt V, Chmielowski B, Evans TRJ, Gastaud L, Linette G, Berking C, Schachter J, Rodrigues MJ, Shoushtari AN, Clemett D, Ghiorghiu D, Mariani G, Spratt S, Lovick S, Barker P, Kilgour E, Lai Z, Schwartz GK, Nathan P. Selumetinib in Combination With Dacarbazine in Patients With Metastatic Uveal Melanoma: A Phase III, Multicenter, Randomized Trial (SUMIT). J Clin Oncol. 2018 Apr 20;36(12):1232-1239. doi: 10.1200/JCO.2017.74.1090. Epub 2018 Mar 12. PMID 29528792